CLINICAL TRIAL: NCT01031719
Title: A Phase III, Randomized, Controlled, Open Label Study to Evaluate the Immunogenicity, Safety, and Tolerability of an Adjuvanted A(H1N1) Vaccine Versus Non-Adjuvanted Vaccines Against Novel H1N1 Virus in Patients With Invasive Solid Tumors
Brief Title: Clinical Trial to Compare the Immunogenicity, Safety, and Tolerability of an Adjuvanted A(H1N1) Influenza Vaccine Versus Non-Adjuvanted A(H1N1) Influenza Vaccines in Patients With Invasive Solid Tumors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiltern Pesquisa Clinica Ltda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V111_15TP
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: H1N1 Influenza Virus; Invasive Solid Tumors
Keywords: Influenza A Virus; Virus Diseases; Influenza, Human; H1N1; Immunogenicity; safety; tolerability; tumors; oncology
MeSH Terms: conditions — Virus Diseases; Influenza, Human; Neoplasms | interventions — Influenza Vaccines

ARMS (4):
- Group A: High Risk Population (Experimental): Each subject will receive two doses of the assigned vaccine, the first on Study Day 1, and the second on Study Day 22
  Interventions: Biological: adjuvanted A(H1N1) influenza vaccine
- Group B: High Risk Subjects (Experimental): Each subject will receive two doses of the assigned vaccine, the first on Study Day 1, and the second on Study Day 22
  Interventions: Biological: non-adjuvanted A(H1N1) influenza vaccine
- Group C: Healthy Subjects (Experimental): Each subject will receive two doses of the assigned vaccine, the first on Study Day 1, and the second on Study Day 22
  Interventions: Biological: adjuvanted A(H1N1) influenza vaccine
- Group D: Healthy Subjects (Experimental): Each subject will receive two doses of the assigned vaccine, the first on Study Day 1, and the second on Study Day 22
  Interventions: Biological: non-adjuvanted A(H1N1) influenza vaccine

INTERVENTIONS:
Biological: adjuvanted A(H1N1) influenza vaccine — 7.5 ug of HA antigen; adjuvanted; monovalent
  Arms: Group A: High Risk Population; Group C: Healthy Subjects
Biological: non-adjuvanted A(H1N1) influenza vaccine — 15ug of HA antigen, non-adjuvanted; trivalent
  Arms: Group B: High Risk Subjects
Biological: non-adjuvanted A(H1N1) influenza vaccine — 15 mcg of antigen; non-adjuvanted; trivalent
  Arms: Group D: Healthy Subjects

SUMMARY:
This is a phase III, randomized, controlled, open label study with two vaccine regimens. The study will assess the relative safety and immunogenicity of vaccine regimens comparing adjuvanted versus non-adjuvanted formulations of A(H1N1) inactivated influenza virus vaccine in subjects with Solid Invasive Tumors and to compare safety and immunogenicity data with a contemporaneously enrolled control group of age-comparable, healthy subjects.

Because certain individuals may be hypo-responsive to influenza vaccination, additional studies with high-risk groups are warranted in order to determine the optimal vaccine formulation and dosing schedule for prevention of novel H1N1 virus infection.

ELIGIBILITY:
Inclusion Criteria:

For Invasive Solid Tumor Subjects:

* Subjects between 2 and 70 years of age (inclusive)
* Any sex or ethnicity
* Confirmed diagnosis of Invasive Solid Tumor or hematological malignancies in complete remission for at least 3 months and not more than 18 months after the last neo-adjuvant and/or adjuvant chemotherapy cycle according to investigators assessment and the subjects medical records
* Previous use of neo-adjuvant and/or adjuvant chemotherapy for the treatment on an invasive solid tumor
* Life expectancy of at least 12 months
* Karnofsky Performance Scale > 40%
* Childbearing potential women must be willing to use an acceptable contraceptive method. Acceptable contraceptive methods are defined as one or more of the following:

  1. Hormone contraceptive (such as oral, injectable, transdermal patch, subcutaneous implant, cervical ring)
  2. Barrier (condom with spermicide or diaphragm with spermicide) at each intercourse and during the whole intercourse
  3. Intra-uterine device (IUD)
  4. Monogamous relation with vasectomized partner (must have been vasectomized at least six months before the volunteer entered the study).
* Subjects capable of following all the study procedures and available for all visits scheduled to the investigation site
* Subjects capable of understanding the nature and risk of the study proposed and sign the consent form
* In case of children and adolescents (below 18 years of age): Subjects capable of understanding the nature of the study and whose legal guardian understands the nature and risk of the study proposed and signs the consent form
* The study subjects may have other underlying chronic diseases that do not involve immunosuppression (e.g. osteoarticular diseases, cardiorespiratory diseases, metabolic diseases, stable, non progressive, non-severe neurologic disorders without cognitive impairment, ophthalmologic diseases, etc.), but their symptoms/signs must be under control through medical follow-ups and drug therapy

For Healthy Subjects:

* Subjects between 2 and 70 years of age (inclusive)
* Any sex and ethnicity
* Subjects with good health as determined by medical history, physical evaluation, and investigator's clinical opinion
* Childbearing potential women must be willing to use an acceptable contraceptive method. Acceptable contraceptive methods are defined as one or more of the following:

  1. Hormone contraceptive (such as oral, injectable, transdermal patch, subcutaneous implant, cervical ring)
  2. Barrier (condom with spermicide or diaphragm with spermicide) at each intercourse and during the whole sexual intercourse
  3. Intra-uterine device (IUD)
  4. Monogamous relation with vasectomized partner (must have been vasectomized for at least six months before the volunteer entered the study).
* Subjects capable of respecting all the study procedures and available for all the visits scheduled at the investigation site
* Subjects capable of understanding the nature and risk of the study proposed and sign the consent form
* In case of children and adolescents (below 18 years of age): Subjects capable of understanding the nature of the study and whose legal guardian understands the nature and risk of the study proposed and signs the consent form

Exclusion Criteria:

For Invasive Solid Tumor Subjects:

* Previous laboratory confirmed diagnosis of an infection by the novel H1N1 virus
* Administration of other vaccine against the novel H1N1 virus within 3 months prior to inclusion in the study
* Any recent vaccine given within the last 21 days (inclusive)
* History of allergic reaction to an influenza vaccine in the past, or a current or previous occurrence of allergy to egg or egg protein, kanamycin, and neomycin sulfate
* Acute febrile disease (vaccination may be delayed up to 3 days after the resolution of the symptoms)
* Presence of other diseases, not related to cancer with confirmed immunosuppression
* Chemotherapy, biologic therapy or radiation within 3 months prior to inclusion in the study
* History of chronic hepatic or renal disease
* History of cognitive disorders
* History of progressive or severe neurological disorders, including Guillain-Barré Syndrome
* Pregnancy or breast-feeding
* Use of immunomodulatory therapy, including cyclosporin, interleukins, and interferons, within 3 months prior to inclusion in the study
* Receipt of parenteral immunoglobulin, hemotherapy, and/or plasma derivatives within 3 months prior to inclusion in the study
* Receipt of any investigational product within 12 months prior to inclusion in the study

For Healthy Subjects:

* Previous laboratory confirmed diagnosis of an infection by the new virus H1N1
* Receipt of another vaccine against the new virus H1N1 within 3 months prior to inclusion in the study
* Any recent vaccine given within the last 21 days (inclusive)
* History of allergic reaction to influenza vaccine in the past, or a current or previous allergy to egg or egg protein, kanamycin, and neomycin sulfate;
* Acute febrile disease (the vaccination may be delayed up to 3 days after symptoms resolution)
* Pregnancy or breast-feeding
* Receipt of parenteral immunoglobulin, hemotherapy, and/or plasma derivatives within 3 months prior to inclusion in the study;
* Receipt of any investigational product within 12 months prior to inclusion in the study

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2010-08; Primary Completion 2011-09 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to determine the optimal influenza vaccination strategy in patients with invasive solid tumors | 3 months

SECONDARY OUTCOMES:
Assess whether the adjuvanted vaccine offers a meaningful benefit in relation to the non-adjuvanted vaccine in this at-risk population | 3 months
Assess whether two doses of either study vaccine will provide meaningful benefit in comparison to one dose | 3 months
Assess the persistence of antibody levels in the two vaccine groups | 3 months
Gain further insight into the safety of the adjuvanted and non-adjuvanted H1N1 vaccines in this high-risk patient population | 3 months

CONTACTS AND LOCATIONS:
Locations (3):
- Brazil (3):
  - BIOCANCER Clinical Research, Belo Horizonte, Minas Gerais
  - Centro de Estudos e Pesquisas de Oncologia e Hematologia da Faculdade de Medicina da Fundação do ABC, Santo André, São Paulo
  - Universidade Federal de São Paulo, São Paulo, São Paulo

REFERENCES:
- [Background] Clark TW, Pareek M, Hoschler K, Dillon H, Nicholson KG, Groth N, Stephenson I. Trial of 2009 influenza A (H1N1) monovalent MF59-adjuvanted vaccine. N Engl J Med. 2009 Dec 17;361(25):2424-35. doi: 10.1056/NEJMoa0907650. Epub 2009 Sep 10. PMID 19745215
- [Background] Novel Swine-Origin Influenza A (H1N1) Virus Investigation Team; Dawood FS, Jain S, Finelli L, Shaw MW, Lindstrom S, Garten RJ, Gubareva LV, Xu X, Bridges CB, Uyeki TM. Emergence of a novel swine-origin influenza A (H1N1) virus in humans. N Engl J Med. 2009 Jun 18;360(25):2605-15. doi: 10.1056/NEJMoa0903810. Epub 2009 May 7. PMID 19423869
- [Background] Gross PA, Gould AL, Brown AE. Effect of cancer chemotherapy on the immune response to influenza virus vaccine: review of published studies. Rev Infect Dis. 1985 Sep-Oct;7(5):613-8. doi: 10.1093/clinids/7.5.613. PMID 3903940
- [Background] Kunisaki KM, Janoff EN. Influenza in immunosuppressed populations: a review of infection frequency, morbidity, mortality, and vaccine responses. Lancet Infect Dis. 2009 Aug;9(8):493-504. doi: 10.1016/S1473-3099(09)70175-6. PMID 19628174